CLINICAL TRIAL: NCT04826757
Title: Effectiveness of Coordinated Care to Reduce the Risk of Prolonged Disability Among Patients Suffer From Subacute or Recurrent Acute Low Back Pain in Primary Care
Brief Title: Effectiveness of Coordinated Care to Reduce the Prolonged Disability Risk Among Patients Suffering From Low Back Pain in Primary Care
Acronym: COLOMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-A01039-30
Record Dates: First submitted 2021-03-03; First posted 2021-04-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, cluster trial. the project is multicentered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care (No Intervention): standard care for low back pain management by general practioners (GPs). the physiotherapist and occupational health services can be solicited independently by the patient or GP.
- coordinated care (Experimental): Coordinated care between general practioners, physiotherapist and occupational health services.
  An intervention training will be performed before the start of the study for any care professional's to elaborate coordination tools and have an active communication.
  Interventions: Other: Coordinated care

INTERVENTIONS:
Other: Coordinated care — Coordinated care between general practioners; physiotherapists and occupational health services.
  Early contact with occupational health service by the general practioner and use of occupational retention tool Active physiotherapy (Individual active, intensive and regular rehabilitation program with 15 sessions of 1 hour, at a rate of 2 or 3 sessions per week)
  Arms: coordinated care

SUMMARY:
Common low back pain affects about 23% of general population and can be associated with psychosocial difficulties and prolonged inability to work. Its management in France mainly depends on general practioners, and sometime on physiotherapists.

A coordinated care between general practioners, physiotherapists and occupational health services would help to improve the care pathway for patients and health professionals.

The main objective is to assess the impact of coordinated primary care and deployed at the territories' level, in subacute or acute recurrent low back pain patients in comparison with the standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting an investigator GP for subacute low back pain or acute recurrent low back pain
* Patient with occupational activity (including sick leave)
* Patient depending of occupational health service
* Obtaining the signature of the consent to participate in this trial
* Patient Registered with social security scheme

Non-inclusion Criteria:

* Specific low back pain (fracture, infection, osteoporosis, inflammatory disease, tumor)
* Low back pain with sciatic, cruralgia
* Contraindication to active reeducation
* Impossibility to follow up during 12 months
* Patient planning to retire within the 12 months following the enrollment
* Disability to write or read french
* Adult patient protected under the law (guardianship),
* Pregnant, breastfeeding or parturient women
* Persons deprived of their liberty by judicial or administrative decision
* Persons subject to legal protection measures
* Persons unable to consent
* Persons on coercion psychiatric care
* Physiotherapy by a physiotherapist who don't participate in this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Perceived inability at 1 year | Enrollment to 12 months follow up
  Ratio of patient presenting improvement equal or above 4 points of Roland Morris Disability Questionnaire. The minimum value of Roland Morris Disability Questionnaire is 0 and the maximun value is 24. A higher score mean worse outcome

SECONDARY OUTCOMES:
Perceived inability | Enrollment to 3 months follow up, Enrollment to 6 months follow up
  Ratio of patient presenting improvement equal or above 4 points of Roland Morris Disability Questionnaire. The minimum value of Roland Morris Disability Questionnaire is 0 and the maximun value is 24. A higher score mean worse outcome
Roland Morris Disability score over time | Enrollment, 3 months, 6 months, 12 months
  Evolution of Roland Morris Disability Questionnaire over time. The minimum value is 0 and the maximun value is 24. A higher score mean worse outcome
Pain perceived | Enrollment - 3 months , Enrollment - 6 months and Enrollment -12 months
  Ratio of patients presenting improvement equal or above 2 points of numerical pain scale The minimum value is 0 and the maximun value is 10. A higher score mean worse outcome
Numerical pain scale over time | Enrollment, 3 months, 6 months, 12 months
  Evolution of numerical pain scale over time. The minimum value is 0 and the maximun value is 10. A higher score mean worse outcome
Occupational status | at 3 months, 6 months and 12 months
  Ratio of patients having an active occupation (defined by have an employment and be present at work )
Employment rate | Enrollment, 3 months, 6 months, 12 months
  Evolution of employment rate over time
Sick leave | during 12 months after inclusion
  number of sick leave days
Improved patients | at 3 months, 6 months and 12 months
  Ratio of improved patients. Improved patients is defined by patient presenting improvement equal or above 4 points of Roland Morris Disability Questionnaire and improvement equal or above 2 points of numerical pain scale and having a active occupational
Evolution of improved patients ratio | Enrollment, 3 months, 6 months, 12 months
  Evolution of improved patients ratio over time Improved patients is defined by patient presenting improvement equal or above 4 points of Roland Morris Disability Questionnaire and improvement equal or above 2 points of numerical pain scale and having a active occupational
Mental component score of Short Form -12 | Enrollment, 3 months, 6 months, 12 months
  Evolution of mental scores over time The mental component score is determined by 4 categories of Short Form -12. The minimum value of each category is 0 and the maximun value is 100. A higher score mean better outcome
Physical component score of Short Form -12 | Enrollment, 3 months, 6 months, 12 months
  Evolution of physical scores over time. The physical component score is determined by 4 categories of Short Form -12. The minimum value of each category is 0 and the maximun value is 100. A higher score mean better outcome
Occupational component score of Fear Avoidance Beliefs Questionnaire | Enrollment, 3 months, 12 months
  Evolution of occupational component score over time. Occupational component is assessed using the Fear Avoidance Beliefs Questionnaire.
  The minimum value is 0 and the maximun value is 42. A higher score mean worse outcome
Physical activity component score of Fear Avoidance Beliefs Questionnaire | Enrollment, 3 months, 12 months
  Evolution of physical activity component score over time. Physical activity component is assessed using the Fear Avoidance Beliefs Questionnaire.
  The minimum value is 0 and the maximun value is 24. A higher score mean worse outcome
Anxiety component score of Hospital Anxiety and Depression Scale | Enrollment 3 months, 12 months
  Evolution of Anxiety score over time Anxiety Component is assessed using the Hospital Anxiety and Depression Scale The minimum value is 0 and the maximun value is 21. A higher score mean worse outcome
Depression component score of Hospital Anxiety and Depression Scale | Enrollment, 3 months, 12 months
  Evolution of Depression score over time Depression component is assessed using the Hospital Anxiety and Depression Scale The minimum value is 0 and the maximun value is 21. A higher score mean worse outcome
Coordination care score of Patient Centered Coordination by a Care Team questionnaire | Enrollment, 3 months, 12 months
  Evolution of coordination care score over time This score is assessed by using Patient Centered Coordination by a Care Team questionnaire.
  The minimum value is 0 and the maximun value is 42. A higher score mean better outcome
GP satisfaction related to patient care | T0 = baseline (cluster initiation); T1 = 1 year (6 months after inclusion of the 5th cluster patient); T2 = through study completion, an average of 3 years (12 months after the last cluster patient inclusion)
  Evolution of GP satisfaction using an numerical scale The minimum value is 0 and the maximun value is 10. A higher score mean worse outcome
Physiotherapist satisfaction related to patient care | T0 = baseline (cluster initiation); T1 = 1 year (6 months after inclusion of the 5th cluster patient); T2 = through study completion, an average of 3 years (12 months after the last cluster patient inclusion)
  Evolution of physiotherapist satisfaction using an numerical scale The minimum value is 0 and the maximun value is 10. A higher score mean worse outcome
Professionals trained for intervention | Baseline intervention formations
  number of professionals trained for intervention
Biomechanical component score of Pain Attitudes and Beliefs score - for intervention physiotherapists | T0 = baseline (cluster initiation); T1 = 1 year (6 months after inclusion of the 5th cluster patient); T2 = through study completion, an average of 3 years (12 months after the last cluster patient inclusion)
  Evolution of Biomechanical component score for intervention physiotherapists. Biomechanical component is assessed using the Pain Attitudes and Beliefs Score. The minimum value is 10 and the maximun value is 60. A higher score mean worse outcome
Biopsychosocial component score of Pain Attitudes and Beliefs score - for intervention physiotherapists | T0 = baseline (cluster initiation); T1 = 1 year (6 months after inclusion of the 5th cluster patient); T2 = through study completion, an average of 3 years (12 months after the last cluster patient inclusion)
  Evolution of Biopsychosocial component score for intervention physiotherapists. Biopsychosocial component is assessed using the Pain Attitudes and Beliefs Score.The minimum value is 9 and the maximun value is 54. A higher score mean better outcome
Biopsychosocial component score of Pain Attitudes and Beliefs score - for GPs | T0 = baseline (cluster initiation); T1 = 1 year (6 months after inclusion of the 5th cluster patient); T2 = through study completion, an average of 3 years (12 months after the last cluster patient inclusion)
  Evolution of Biopsychosocial component score for GPs. Biopsychosocial component is assessed using the Pain Attitudes and Beliefs Score.The minimum value is 9 and the maximun value is 54. A higher score mean better outcome
Biomechanical component score of Pain Attitudes and Beliefs score - for GPs | T0 = baseline (cluster initiation); T1 = 1 year (6 months after inclusion of the 5th cluster patient); T2 = through study completion, an average of 3 years (12 months after the last cluster patient inclusion)
  Evolution of Biomechanical component score for GPs. Biomechanical component is assessed using the Pain Attitudes and Beliefs Score. The minimum value is 10 and the maximun value is 60. A higher score mean worse outcome
Professional dialogues | during the 12 months of follow up
  Existence and types of dialogues between GP and other professionals
Number of consultations or sessions | during the 12 months of follow up
  Number of consultations or sessions

CONTACTS AND LOCATIONS:
Overall Officials: Aline RAMOND ROQUIN, MD-PHD, Principal Investigator — Department of Family Medicine - University of Angers
Locations (20):
- France (20):
  - Cluster Bonchamp, Bonchamp-lès-Laval
  - Cluster Vaunoise, Breteil
  - Cluster BRULON, Brûlon
  - Cluster Château Gontier, Château-Gontier
  - Cluster Châteauneuf sur Sarthe / Morannes, Châteauneuf-sur-Sarthe
  - Cluster Clisson, Clisson
  - Cluster Conlie, Conlie
  - Cluster Craon Renaze Cosse, Craon
  - Cluster Entrammes Laval, Entrammes
  - Cluster Roche sur Yon, La Roche-sur-Yon
  - Cluster Chantenay, Nantes
  - Cluster Dinan / Quévert / Plouasne, Quévert
  - Cluster Rennes Beauregard, Rennes
  - Cluster Rennes Villejean, Rennes
  - Cluster Les Collines, Roquefort-les-Pins
  - Cluster St Florent, Mauges, Possonnière, Saint-Florent-le-Vieil
  - Cluster Savenay, Savenay
  - Cluster SEGRE, Segré
  - Cluster Angers- Trélazé, Trélazé
  - Cluster Vence, Vence

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).

REFERENCES:
- [Derived] Ramond-Roquin A, Begue C, Vizzini J, Chhor S, Bouchez T, Parot-Schinkel E, Loiez A, Petit A, Ghali M, Peurois M, Bouton C. Effectiveness of coordinated care to reduce the risk of prolonged disability among patients suffering from subacute or recurrent acute low back pain in primary care: protocol of the CO.LOMB cluster-randomized, controlled study. Front Med (Lausanne). 2023 Jun 20;10:1156482. doi: 10.3389/fmed.2023.1156482. eCollection 2023. PMID 37409270